CLINICAL TRIAL: NCT03851471
Title: An Open-label, Single-institution, Non-randomized, Single-arm, Pilot Study of Jiu-wei-zhen-xiao Granule for the Treatment in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Jiu-wei-zhen-xiao Granule for Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhong Wang (Other)
Responsible Party: Sponsor-Investigator, Zhong Wang, Vice-director, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JIUWEI-Gan 1-Ver1.0
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jiu-wei-zhen-xiao Granule (Experimental): Patients will be treated for 12 weeks, with oral administration of 5g once of Jiu-wei-zhen-xiao Granule,three times a day, based on the conventional treatment for HCC, such as antiviral treatment, supportive treatment or symptomatic treatment.
  Interventions: Drug: Jiu-wei-zhen-xiao Granule

INTERVENTIONS:
Drug: Jiu-wei-zhen-xiao Granule — Patients will be treated for 12 weeks, with oral administration of 5g once of Jiu-wei-zhen-xiao Granule,three times a day, based on the conventional treatment for HCC, such as antiviral treatment, supportive treatment or symptomatic treatment.

SUMMARY:
This is a piolt single-arm trial of Jiu-wei-zhen-xiao Granule, extracted from nine kinds of Chinese medicnie, for the treatment in patients with advanced, unresectable hepatocellular carcinoma(HCC). The primary objective is to assess its therapeutic efficacy in patients with unresectable HCC. The primary endpoint is overall survival (OS) after the use of 12-week drug. Secondary endpoints include progression-free survival (PFS) after the use of 12-week drug, the improvement of the score of the European Organization for Reasearch and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30), the changes of the liver function, coagulation function, the size of solid tumors,"Du-tan-yu-jie Zheng" in Chinese medicine, pain Visual Analogue Scale and toxicity profile of Jiu-wei-zhen-xiao Granule.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18~75 years;
2. Patients must have diagnosis of advanced hepatocellular cancer (HCC) by one of the following:

(1) Histopathology; (2) Elevated serum alpha-fetoprotein (AFP) >400 ng/ml and findings on magnetic resonance imaging (MRI) or computed tomography (CT) scans characteristic of HCC; (3) Findings on triple phase MRI or CT scans characteristic of HCC in patients with cirrhosis and tumors at least 1 cm or greater, without a curative treatment option (transplant, resection, or ablation).

3.The clinical staging of HCC is B or C or D staging as the Barceln Clinical Liver Cancer Classification(BCLC);

4. Patients with hepatitis B virus infection;

5. Patients with "Du-tan-yu-jie Zheng" in Chinese medicine;

6. Karnofsky score ≥60;

7. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with unstable vital signs;
2. Any uncontrolled, severe, intercurrent illness including but not limited to ongoing or active infection, heart, brain, lung and other systemic diseases or other kinds of tumors;
3. Known history of allergy to the ingredients of this product;
4. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial through 120 days after the last dose of trial treatment;
5. Receipt of any other investigational agents ≤ 1 month of the first dose of study treatment;
6. Patients who cannot take oral medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-07 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Up to 12 weeks
  Overall Survival (OS) is defined as the percentage of people in a group who are alive after the 12-week use of drug.

SECONDARY OUTCOMES:
Progression-Free Survival | Baseline, 4 weeks, 8 weeks, 12 weeks
  Progression-free survival (PFS) will be defined as the elapsed time from the first date of study treatment until documented disease progression (as per RECIST 1.1) or death from any cause, whichever is earlier. For patients who remain alive without progression, follow-up time will be censored at the date of last disease assessment .
European Organization for Reasearch and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) (Chinese version, Version 3.0) | Baseline, 4 weeks, 8 weeks, 12 weeks
  EORTC QLQ-C30 is a 30-item questionnaire composed of multi-item scales and single items that reflect the multidimensionality of the QoL construct. It includes five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea/vomiting), and a global health status/QoL scale. The remaining single items assess additional symptoms commonly reported by cancer patients (dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea), as well as the perceived financial impact of the disease and treatment.
The level of the liver function | Baseline, 4 weeks, 8 weeks, 12 weeks
  The biochemical indicators of the liver function include alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin(TBiL), direct bilirubin (DBiL), albumin (ALB), alkaline phosphatase (AKP), gamma-Glutamyltransferase (γ-GGT).
The level of AFP | Baseline, 4 weeks, 8 weeks, 12 weeks
  AFP is the abbreviation of alpha fetoprotein, which could be the progress of the primary hepatocellular carcinoma
The level of coagulation function | Baseline, 12 weeks
  The biochemical indicators of the coagulation function include prothrombin time (PT), activated partial thromboplastin time (APTT), thrombin time (TT), fibrinogen (FIB).
The size of solid tumors | Baseline, 12 weeks
  The size of solid tumors is measured by a professional film reader using MRI/CT.
"Du-tan-yu-jie Zheng" symptoms score in Chinese medicine | Baseline, 4 weeks, 8 weeks, 12 weeks
  "Du-tan-yu-jie Zheng" is a series of common symptoms in HCC，including distending pain in the hypochondrium,jaundice, a lump below the costal region,weak and lassitude, poor appetite,abdominal distension and fullness,dizziness and tinnitus, bitter or dry mouth,constipation, urinary yellow,upset and irritable,red or dark red tongue, stringy or rapid pulse
10cm-VAS of the pain | Baseline, 4 weeks, 8 weeks, 12 weeks
  The 10cm Visual Analogue Scale (VAS) of the pain is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10) .

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei Provincial Hospital of Traditional Chinese Medicine, Wuhan, Hubei, China